CLINICAL TRIAL: NCT02126995
Title: A 6-week, Randomized, Multicenter, Double-blind, Parallel, Flexed and Fixed-dose Study of MG01CI (Metadoxine Extended-release) Low Dose and High Dose Compared With Placebo in Adults and Adolescents With Fragile X Syndrome
Brief Title: A 6-week, Study of MG01CI Low Dose and High Dose Compared With Placebo in Adults and Adolescents With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL014
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2014-12

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome, Fra(X) Syndrome, FRAXA Syndrome
MeSH Terms: conditions — Fragile X Syndrome; Syndrome | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metadoxine Immediate/Slow-release (Experimental): Flexed and fixed-dose Metadoxine Immediate/Slow-release 700 mg and 1400 mg administered orally once daily
  Interventions: Drug: MG01CI extended-release tablet
- Placebo (Placebo Comparator): Placebo tablet identical in appearance to study investigational product. Administered orally once daily
  Interventions: Drug: MG01CI extended-release tablet

INTERVENTIONS:
Drug: MG01CI extended-release tablet — Metadoxine, MG01CI extended-release tablet taken for 6 weeks treatment. Starting with a dose of 700 mg for 2 weeks followed by a 2 weeks of 1400 mg and then 2 weeks of 700 mg or 1400 mg.
  Other Names: Metadoxine (pyridoxol L-2-pyrrolidone-5-carboxylate)

SUMMARY:
This study is a multisite, randomized, double-blind, placebo-controlled, phase 2 study of MG01CI (low dose and high dose once daily) for 6 weeks compared with placebo in a 1:1 ratio of 60 adolescent and adult subjects with Fragile X Syndrome (FXS). Following Screening, subjects will be randomized to MG01CI or matching placebo at Baseline (Day 0) and the 6 week Double-blind Treatment Period will begin on Day 1.

The first 4 weeks of the treatment period will be a dose-optimization period,

All subjects will start with two daily tablets: low dose metadoxine or matching blinded placebo. At weekly visits/phone assessments, the investigator will evaluate the dose based upon the investigator's assessment of safety and tolerability. If the subject demonstrates safety or tolerability concerns with the low dose after 1 or 2 weeks of treatment, then the subject will be discontinued. If there are no concerns about safety and tolerability after 2 weeks of treatment, then the dose will be increased to high dose or placebo. If at the high dose there are concerns about safety and tolerability, then the dose will be either kept the same or reduced to low dose for the remainder of the treatment period.

There will be a 2-week Follow-up Period after the last dose of study treatment or early termination.

DETAILED DESCRIPTION:
This study is a multisite, randomized, double-blind, placebo-controlled, phase 2 study of MG01CI (low and high doses of metadoxine once daily) for 6 weeks compared with placebo in a 1:1 ratio of 60 adolescent and adult subjects with FXS. Following Screening, subjects will be randomized to MG01CI or matching placebo at Baseline (Day 0) and the 6 week Double-blind Treatment Period will begin on Day 1.

The first 4 weeks of the treatment period will be a dose-optimization period, during which the subject's dose of MG01CI or placebo will be optimized. Investigators and subjects will be blinded with regard to whether the subject is taking active drug or placebo. Subjects will be blinded to anticipated dose (low vs high dose), while Investigators will not be blinded to anticipated dose, low dose vs high dose. Every two weeks subjects will receive 2-week supply treatment. A phone follow-up assessment of safety and tolerability will occur during titration after 1 and 3 weeks of treatment; if the investigator has any significant concerns regarding safety and tolerability, the subject will be assessed at the site at an unscheduled visit. All subjects will be assessed at the site after 2 weeks and 4 weeks of treatment.

All subjects will start with either low dose or matching blinded placebo (2 tablets daily). At weekly visits/phone assessments, the investigator will evaluate the dose based upon the investigator's assessment of safety and tolerability. If the subject demonstrates safety or tolerability concerns with the low dose after 1 or 2 weeks of treatment, then the subject will be discontinued. If there are no concerns about safety and tolerability after 2 weeks of treatment, then the dose will be increased to 2 tablets of either high dose of active treatment or placebo. If at high dose there are concerns about safety and tolerability, then the dose will be either kept the same or reduced to low dose for the remainder of the treatment period.

The last 2 weeks of the treatment period will be a dose-maintenance period. During the dose-maintenance period, the subject will maintain his or her optimal dose as determined at the end of the dose-optimization period. A phone follow-up assessment of safety and tolerability will occur after 5 weeks of treatment (after 1 week of dose maintenance). If the investigator has any significant concerns regarding safety and tolerability, the subject will be assessed at the site at an unscheduled visit. The subject will be assessed at the site after 6 weeks of treatment (after 2 weeks of dose maintenance).

There will be a 2-week Follow-up Period after the last dose of study treatment or early termination.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or a non-pregnant, non-lactating woman aged 15 to 55 years, inclusive, at the Randomization Visit.
2. Subject has Fragile X Syndrome with a molecular genetic confirmation of the full Fragile X Mental Retardation (FMR1) mutation (≥200 CGG repetitions).
3. Subject has a score of 12 or greater on the inattentive subscale of the ADHD RS IV (as rated by the investigator in a clinical interview of the parent/legal authorized guardian/consistent caregiver).
4. Current treatment with no more than 3 prescribed psychotropic medications. Anti epileptic medications are permitted and are not counted as psychotropic medications if they are used for treatment of seizures. Anti-epileptics for other indications, such as the treatment of mood disorders, count towards the limit of permitted medications.

   1. Permitted concomitant psychotropic medications (except anti-epileptic medications and stimulants; see 4b and 4d) must be at a stable dose and dosing regimen for at least 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
   2. Anti-epileptic medications must be at a stable dose and dosing regimen for 12 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
   3. Subjects with a history of seizure disorder who are currently receiving treatment with anti-epileptics must have been seizure-free for 3 months preceding Screening, or must be seizure-free for 3 years if not currently receiving anti-epileptics.
   4. Stimulant medications must be at a stable dose and dosing regimen for 12 weeks prior to Screening and must remain stable during the period between Screening and the end of the treatment period (Week 6/early termination), unless the subject is washing out; see Exclusion Criterion 4.
5. Behavioral treatments (excluding psychotherapy; see exclusion criteria) must be stable for 4 weeks prior to Screening and must remain stable during the period between Screening and the commencement of study medication.
6. Subject has a parent, legal authorized guardian or consistent caregiver who interacts with the subject for at least 10 hours per week and is able to provide weekly rating forms of the subject's behavior.
7. Male and Female subjects of childbearing potential must agree to use an effective contraceptive throughout the study (eg, oral contraceptives or Norplant®; a reliable double barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam]; intrauterine devices; vasectomy; or abstinence) and for at least a month after the study, and females must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit. Females of childbearing potential are defined as women who are between menarche and 2 years post-menopause and who are not surgically sterilized. Male and female subjects who are not sexually active, and who agree to be abstinent throughout the study, will not be required to use birth control.
8. Subject and caregiver are able to attend the clinic regularly and reliably.
9. Subject is able to swallow tablets and capsules.
10. For subjects who are not their own legal guardian, subject's parent/legal authorized guardian is able to understand, read, write, and speak English fluently to complete the study-related materials (or Hebrew for Israeli subjects).
11. For subjects who are not their own legal guardian, subject's parent/legal authorized guardian is able to understand and sign an informed consent form to participate in the study.
12. If subject is his/her own legal guardian, he/she can understand and sign informed consent to participate in the study.
13. If subject is not their own legal guardian, the subject provides assent for participation in the study, if the subject has the cognitive ability to provide assent

Exclusion Criteria:

1. Treatment within the 2 weeks prior to randomization (and throughout the clinical trial) with lithium, acamprosate, racemic baclofen, investigational metabotropic glutamate receptor subtype 5 (mGluR5) medications, d-cycloserine, oxytocin, carbetocin, modafinil, armodafinil, benzodiazepines (unless used for seizure control), memantine, amantadine, bupropion, or any medication in the statin class.
2. Treatment within the 2 weeks prior to Screening with monoamine oxidase (MAO) inhibitors, tricyclic antidepressants, l-dopa, cisplatin, phenobarbital or phenytoin.
3. Current treatment with an N-methyl-D-aspartate (NMDA) antagonist.
4. While stimulants will not be excluded from the trial, the subject and the parent/legal authorized guardian may decide to stop stimulant medication prior to the study upon discussion with the investigator at the Screening visit. If stimulant medication is stopped at screening, a two-week washout is required. A subject that decides to washout from stimulants will be excluded from the trial if a stimulant is administered after the Screening visit or during the course of the trial.
5. Subject is planning to commence psychotherapy or cognitive behavior therapy (CBT) during the period of the study or had begun psychotherapy or CBT within 6 weeks prior to Screening.

   1. A subject who started psychotherapy or CBT for the first time within 6 weeks prior to Screening is excluded.
   2. If a subject was previously receiving psychotherapy or CBT, and is resuming the therapy (such as return from summer vacation), then the subject is eligible for the study if the same therapy was resumed at least 2 weeks before screening.
6. History of or current cardiovascular, renal, hepatic, respiratory, or gastrointestinal disease that may interfere with the absorption, distribution, metabolism, or excretion of the study medication, or that may interfere with the interpretation of the safety, tolerability, or efficacy of the study medication.
7. History of or current cerebrovascular disease or clinically significant brain trauma.
8. Current major depressive disorder (subject must be free of the most recent episode for 3 months prior to randomization).
9. History of a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)-defined substance use disorder in the 3 months prior to Screening.
10. Clinically significant abnormalities, in the investigator's judgment, in safety laboratory tests, vital signs, or ECG, as measured at Screening.
11. Significant hearing or visual impairment that may affect the subject's ability to complete the test procedures.
12. Enrollment in another clinical trial within the 30 days preceding Screening.
13. Any psychiatric condition (eg, schizophrenia or personality disorder as diagnosed by DSM-IV) or clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation as determined by the investigator using medical history, physical examination, neurological examination, laboratory tests, and electrocardiograms. Common diseases such as mild hypertension, well-controlled type 2 diabetes mellitus (hemoglobin A1C [Hgb A1C] <6.5%), etc. are allowed per the investigator's judgment as long as they are stable and controlled by medical therapy that is constant for at least 8 weeks before randomization and subsequently throughout the study. If there are any concerns about the suitability of the subject's medical or surgical condition, the investigator should review the subject's history with the medical monitor. Subjects with autism spectrum disorder or anxiety disorder will be allowed.
14. Subject has known or suspected human immune deficiency virus-positive status or has diseases such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
15. Subject has a history of an allergy or sensitivity to B-complex vitamins.
16. Subject has used mega-dose vitamin B6/pyridoxine during the 28 days before the Randomization Visit. Subjects will be allowed to have a 28-day washout of mega-dose vitamin B6/pyridoxine after the Screening visit. Routine multivitamin supplements will be allowed.
17. Subject has used high-dose supplements of omega-3 fatty acids ≥ 500 mg (such as softgels, capsules, or fish oils; regular daily dietary consumption of fish is allowed) or folic acid supplements (other than routine multivitamin supplements) at any time during the 2 weeks before the Randomization Visit.
18. Subject is related to anyone employed by the sponsor, investigator, or study staff.
19. Subject has any condition that, in the principal investigator's opinion, would place the subject at risk or influence the conduct of the study or interpretation of results.
20. Subject is pregnant, lactating, or using an inadequate contraceptive method. -

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of MG01CI by Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale (ADHD RS-IV) | 6 weeks
  To evaluate the efficacy of MG01CI (Metadoxine Extended-release) once daily compared with placebo in the treatment of symptoms of FXS in adults and adolescents as measured by the inattentive subscale of the Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale (ADHD RS-IV) (as rated by the investigator in a clinical interview of the parent/legal authorized guardian/consistent caregiver).

SECONDARY OUTCOMES:
Evaluation of efficacy of MG01C as measured by total score on the ADHD RS-IV. | 6 weeks
  To evaluate the efficacy of MG01CI (Metadoxine Extended-release) once daily compared with placebo in the treatment of symptoms of FXS in adults and adolescents as measured by the total score on the ADHD RS-IV.

OTHER OUTCOMES:
Evaluation of safety by AE's count | 6 weeks
  To evaluate the safety, and tolerability of treatment with MG01CI once daily on the adverse events (AEs);
Evaluation of safety by AE's vital sign measurements | 6 weeks
Safety evaluation by lab tests (hematology, chemistry, and urinalysis) | 6 weeks
Evaluation of safety by physical and neurological examinations | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (12):
- United States (11):
  - Southwest Autism Research & Resource Center, Phoenix, Arizona
  - University of California Davis Pediatrics, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - RUSH University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Baylor College of Medicine Research, Houston, Texas
  - Univ. of Washington/Seattle Children's Hospital, Seattle, Washington
- Sheba Academic Medical Center, Ramat Gan, Israel, Israel